CLINICAL TRIAL: NCT05149547
Title: The Comparison of mNGS Versus Blood Culture for Early Diagnosis of Blood Stream Infection During the Febrile Neutropenia in Patients With Hematological Disease
Brief Title: mNGS Versus Blood Culture in FN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University International Hospital (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Head of Peking University Institute of Hematology, Peking University People's Hospital
Other Study IDs: mNGS for FN(2021PHB362-001)
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Infections; Hematologic Diseases; Febrile Neutropenia
MeSH Terms: conditions — Infections; Hematologic Diseases; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood culture versus mNGS detection — peripheral 4ml for mNGS detection

SUMMARY:
Blood stream infection (BSI) during febrile neutropenia (FN) is a lethal complication, while confirmed diagnosis via blood culture is usually with low sensitivity and time delay. The new technique of metagenome next generation sequencing (mNGS) has the potential of early and more accurate detection of pathogens. However, this technique has not been well validated for BSI diagnosis in patients with hematological disease. Therefore, we designed a prospective multicenter study to compare the diagnosis performance in BSI.

ELIGIBILITY:
Inclusion Criteria:

* hematologic disease
* febrile neutropenia

Exclusion Criteria:

* refuse to consent
* age<=14
* not caused by infection

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with hematologic disease during febrile neutropenia
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
diagnosis performance | 14 days after sapmpling
  the sensitivity and specificity of mNGS

CONTACTS AND LOCATIONS:
Overall Officials: YUQIAN SUN, MD, Principal Investigator — Peiking University People's Hospital
Locations (1):
- Yuqian Sun, Beijing, China

IPD SHARING:
Plan to Share IPD: No